CLINICAL TRIAL: NCT03064243
Title: Effectiveness and Safety of Apatinib for the Patients With Advanced Soft Tissue Sarcoma
Brief Title: A Phase II Study of Apatinib in STS Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Yao, Professor, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-S301
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib group (Experimental): apatinib 500mg po qd
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — apatinib 500mg po. qd.
  Other Names: apatinib mesylate tablets

SUMMARY:
Apatinib is a kind of innovative medicines approved by China Food and Drug Administration（CFDA）, which was researched by Jiangsu Hengrui Pharmaceutical Co., Ltd. Apatinib is a kinase inhibitor of receptor tyrosine with VEGFR2. The protocol is to explore Apatinib for the effectiveness of advanced soft tissue sarcoma and safety.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologically proven advanced soft tissue sarcoma, At least one measurable lesion. Including: Synovial sarcoma, leiomyosarcoma, Alveolar soft part sarcoma, Undifferentiated pleomorphic sarcoma / malignant fibrous histiocytoma, Liposarcoma, Fibrosarcoma, Clear cell sarcoma, Epithelioid sarcoma, Angiosarcoma, Spindle cell sarcoma, rhabdomyosarcoma treated by chemotherapy, Ewing's sarcoma of soft tissue/Primitive neuroectodermal tumor. Excluding: Malignant peripheral nerve sheath tumor, chondrosarcoma, Dermatofibrosarcoma protuberans, Gastrointestinal stromal tumor, Inflammatory myofibroblastic sarcoma, Malignant mesothelioma.
* Must have evidence of unresectable residual disease.
* In the last 6 months, at least one chemotherapy regimen (including anthracyclines) was used in patients who failed or were unable to tolerate treatment.
* ECOG ps≤2.
* Life expectancy: more than 3 months.
* Prior aptinib less than 2 weeks and at least 1 month since prior aptinib；at least 1 month since prior inhibitor of mTOR or EGFR pathway.
* Not pregnant or nursing；Fertile patients must use effective contraception.
* Hematopoietic

  * HB≥90g/L
  * Absolute neutrophil count ≥ 1,500/mm^3
  * Platelet count ≥ 80,000/mm^3

Exclusion Criteria:

* Uncontrollable hypertension;
* Has influence of oral drugs;
* Patients with high risk of gastrointestinal blooding;
* INR>1.5×ULN，APTT>1.5×ULN;
* Allergic to any ingredient of this product;
* Less than 1 month since last major surgery;
* Brain metastases;
* With the second cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
6 months PFS rate | From baseline to 6 months
  Analyse PFS rate at 6 months

REFERENCES:
- [Derived] Yu W, Zhang H, Chen J, Zhang X, Chen Y, Qu G, Huang G, Zhou Y, Ye T, Fan Z, Yao Y. Efficacy and safety of apatinib in patients with untreated or chemotherapy-refractory soft tissue sarcoma: a multicenter, phase 2 trial. Ann Transl Med. 2022 Sep;10(18):981. doi: 10.21037/atm-22-4229. PMID 36267741